CLINICAL TRIAL: NCT00069017
Title: A Phase II, Randomized, Double-Blind Study to Evaluate the Effects of MEDI-522, a Humanized MAb to Integrin Alpha V Beta 3, On Disease Activity and Progression of Joint Damage in Pts With Active Rheumatoid Arthritis Suboptimally Responding to Methotrexate
Brief Title: Effects of MEDI-522 On Disease Activity and Progression of Joint Damage in Patients With Active Rheumatoid Arthritis Suboptimally Responding to Methotrexate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MI-CP100
Record Dates: First submitted 2003-09-12; First posted 2003-09-17 (Estimated); Last update posted 2007-11-27 (Estimated); Status verified 2007-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — etaracizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Active Comparator): MEDI-522 - 4 mg/kg of MEDI-522 (N=200)
  Interventions: Biological: MEDI-522
- 2 (Placebo Comparator): Placebo (N=100)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: MEDI-522 — MEDI-522 is formulated in a sterile isotonic solution of 10 mM histidine-HCl at pH 6 containing 100 mg of MEDI-522 protein at a concentration of 100 mg/mL.
  Arms: 1
Other: Placebo — Placebo for MEDI-522 contains 10 mM histidine-HCl at pH 6, 0.1% Tween-80, 1.5% Mannitol, 4.3 µg/mL Vitamin B12, and 2 µg/mL D&C Yellow #10.
  Arms: 2

SUMMARY:
To compare, as a preliminary analysis, the effects of MEDI-522 versus placebo at 6 months on disease activity (ACR20) and progression of structural joint damage.

DETAILED DESCRIPTION:
To compare, as a preliminary analysis, the effects of subcutaneously administered MEDI-522 versus placebo at 6 months on disease activity and progression of structural joint damage in patients with rheumatoid arthritis (RA), who have active disease despite ongoing treatment with methotrexate (MTX) with or without hydroxychloroquine (HCQ) and/or sulfasalazine (SSZ).

ELIGIBILITY:
Patients must meet all of the following criteria:

1. Age greater than or equal to 18 (reached 18th birthday or later) at the time of the first dose of study drug
2. Written informed consent obtained from the patient
3. Sexually active females, unless surgically sterile or at least one year post-menopausal, must use an effective method of avoiding pregnancy (including oral, transdermal, injectable, or implanted contraceptives, IUD, female condom, diaphragm with spermicide, cervical cap, abstinence, use of a condom by the sexual partner or sterile sexual partner) for 21 days prior to the first dose of study drug, and must agree to continue using such precautions through 3 months after their last dose of study drug. Cessation of birth control after this point should be discussed with a responsible physician.
4. A diagnosis of RA as defined by American College of Rheumatology (ACR) criteria, which is currently active, as defined by the presence of at least 6 swollen and 6 tender joints involving the hands, wrists, elbows, knees, ankles, or feet and a CRP and/or ESR>Upper Limits of Normal (ULN).
5. Treatment with a stable dose level and frequency of methotrexate for at least 8 weeks prior to study randomization. The patients may also be taking hydroxychloroquine and/or sulfasalazine concurrently with methotrexate. These drugs must also be at stable dose levels and frequencies for at least 8 weeks prior to randomization. Patients currently receiving treatment with stable doses of nonsteroidal anti-inflammatory drugs (NSAIDs), including COX-2 inhibitors, or prednisone (less than or equal to 10 mg/day) will be permitted to continue these medications. Analgesics, including acetaminophen, talwin, propoxyphene, tramadol hydrochloride, codeine or codeine with acetaminophen, hydrocodone, oxycontin, and related medications, will also be permitted. All of these drugs must be at stable dose levels and frequencies for at least 4 weeks prior to study randomization.
6. Prior to randomization (must be within 21 days of the first administration of the study drug), all of the following: WBC ≥ 3,800/mm³; platelet count ≥140,000/mm³; AST, ALT, BUN, or creatinine<1.5 x ULN; stool negative for occult blood; and thyroxine (T4) within normal limits. (Patients with an elevated T4 but with both free T4 and TSH levels within normal limits may be eligible after review by the MedImmune medical monitor.)
7. Willing to forego other forms of experimental treatment during study through Study Day 364
8. Able and willing to complete assessment questionnaires.
9. Willing to participate in study through Study Day 413.

Exclusion Criteria

Patients must have none of the following:

1. Severe active RA, which in the opinion of the investigator currently requires an alternative form of therapy
2. Acute illness at the start of the study
3. Evidence of significant active infection, such as fever greater than or equal to 38.0°C (100.5°F)
4. Known or suspected infection with human immunodeficiency virus (HIV) or other evidence of clinically significant immune deficiencies
5. Evidence of active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection, such as positive HBsAg or positive anti-hepatitis C antibody
6. Insulin-dependent diabetes mellitus that is recent-onset or unstable
7. Evidence of active or latent tuberculosis, which may include a positive PPD skin test result (greater than or equal to 10 mm induration), unless appropriate INH prophylaxis for tuberculosis previously given; a chest X-ray possibly consistent with tuberculosis; or household contact with a patient with active tuberculosis
8. A medical history or evidence of clinically important chronic infection, recurrent (3 or more) infections in the past 6 months requiring antibiotics, or an infection in the past month requiring systemic antibiotics
9. Receipt of any investigational drug therapy, except MEDI-522, within 3 months prior to study randomization (use of licensed agents for indications not listed in the package insert is permitted)
10. Current or any past therapy with anti-TNF biologic antagonists including etanercept, infliximab, and adalimumab
11. Current therapy with cyclosporin A, leflunomide, cyclophosphamide, azathioprine, gold salts, d-penicillamine, mycophenylate mofetil, minocycline or anakinra. These drugs must have been discontinued at least 4 weeks prior to study randomization.
12. Prednisone or equivalent at >10 mg per day orally in the 8 weeks before study randomization. Intraarticular, periarticular, or other forms of parenteral injection of corticosteroids are also not permitted in the 8 weeks prior to study randomization.
13. History of allergic disease or reactions likely to be exacerbated by any component of MEDI-522
14. History of gastrointestinal bleeding (i.e., stool positive for occult blood or overt bleeding) within the previous 6 months
15. Known bleeding disorder or significant risk of clinically important abnormal bleeding due to anticoagulant therapy with warfarin or heparin
16. Elective surgery planned during the study period through Study Day 413
17. Cardiovascular disease that is unstable, such as recent-onset angina, or angina with increasing frequency or severity, or recent myocardial infarction (within past 1 year without definitive corrective surgery such as coronary bypass graft or angioplasty)
18. Neurological disease, such as multiple sclerosis, previous stroke, clinically significant cerebrovascular disease, or other forms of organic brain disease that is clinically significant
19. Pulmonary, hepatic, renal, or hematological disease that is unstable and progressive, or clinically severe
20. Pregnancy (all females, unless surgically sterile or at least one year post-menopausal, must have a negative urine pregnancy test on Study Day 0, prior to dosing)
21. Nursing mother
22. History of alcohol or drug abuse within past 2 years
23. Evidence on physical examination of rheumatoid or other types of vasculitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2003-09; Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (40):
- United States (29):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Sun Valley Arthritis Center, Glendale, Arizona
  - Arizona Research & Education, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - Fayetteville Diagnostic Clinic, Ltd., Fayetteville, Arkansas
  - Thornton Hospital, La Jolla, California
  - Boling Clinical Trials, Rancho Cucamonga, California
  - Pacific Arthritis Center Medical Group, Santa Maria, California
  - Arthritis and Rheumatic Disease Specialty, Aventura, Florida
  - Centre for Rheumatology, Immunology & Arthritis, Fort Lauderdale, Florida
  - Ocala Rheumatology Research Center, Ocala, Florida
  - Sarasota Arthritis Research Center, Sarasota, Florida
  - Sanford S. Hartman, Decatur, Georgia
  - Center for Rheumatology and Bone Research, Wheaton, Maryland
  - RIMA, St Louis, Missouri
  - Arthritis Consultants, Inc., St Louis, Missouri
  - Rheumatology Associates of New Jersey, Teaneck, New Jersey
  - The Center for Rheumatology, Albany, New York
  - Health Research Institute, Oklahoma City, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Oklahoma Center for Arthritis Therapy and Research Inc., Tulsa, Oklahoma
  - Amarillo Center for Clinical Research, Amarillo, Texas
  - Radiant Research, Dallas, Texas
  - Arthritis & Osteoporosis Associates, LLP, Lubbock, Texas
  - University of Utah Medical Hospital, Salt Lake City, Utah
  - The Physician's Clinic of Spokane, Spokane, Washington
  - Rheumatology Northwest/Clinical Trials Northwest, Yakima, Washington
  - Gundersen Clinic Ltd., La Crosse, Wisconsin
  - University of Wisconsin Hospital & Clinics, Madison, Wisconsin
- Canada (11):
  - Richmond Health Science Center, Richmond, British Columbia
  - Manitoba Clinic, Winnipeg, Manitoba
  - Arthritis Centre, Winnipeg, Manitoba
  - Centre Inflammatory Arthritis Disease Studies, Winnipeg, Manitoba
  - Charlton Medical Center, Hamilton, Ontario
  - MAC Research, Inc., Hamilton, Ontario
  - K-W Musculoskeletal Research, Inc., Kitchener, Ontario
  - The Arthritis Program Research Group Inc., Newmarket, Ontario
  - Ottawa General Hospital, Ottawa, Ontario
  - Rheumatic Disease Center of Montreal, Montreal, Quebec
  - Midtown Medical Center, Saskatoon, Saskatchewan